CLINICAL TRIAL: NCT04390984
Title: A Multi-center, Open-label, Fixed-sequence Study of Effect of Gefitinib on the Pharmacokinetics of Apatinib Mesylate in Non-squamous, Non-small-cell Lung Cancer Patients
Brief Title: Drug-drug Interaction Study of Gefitinb on Apatinib in NSCLC Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HR-APTN-DDI-004
Record Dates: First submitted 2020-05-13; First posted 2020-05-18 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: NSCLC
MeSH Terms: interventions — apatinib; Gefitinib

STUDY DESIGN:
Intervention Model Description: All the subjects will administrated with apatinib and gefitinib following the same sequence to assess the effect of gefitinib on the pharmacokinetics of apatinib in NSCLC patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): Subjects will be administrated with 500mg apatinib on day 1 and day 12-15, and administrated with gefitinib on day 4-15.
  Interventions: Drug: Apatinib Mesylate, Gefitinib

INTERVENTIONS:
Drug: Apatinib Mesylate, Gefitinib — Subjects will be administrated with 500mg apatinib on day 1 and day 12-15, and administrated with gefitinib on day 4-15.

SUMMARY:
The primary objective of the study was to assess the effect of gefitinib on the pharmacokinetics of apatinib mesylate in lung cancer patients.

The secondary objective of the study was to assess the pharmacokinetics of gefitinib, and to assess the safety of apatinib mesylate and gefitinib administered in lung cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years of age.
2. ECOG performance status: level 0~1;
3. Anticipated life expectancy ≥ 12 weeks;
4. Lung cancer patients;
5. Major organs in good function;
6. Agree to take approved method of contraception during the clinical trail and 8 weeks after the last dose of apatinib. Female subject should be negative in the pregnancy test;
7. Able to comprehend and willing to sign an informed consent form (ICF)

Exclusion Criteria:

1. History of drug allergy, or allergic to apatinib or gefitinib or ingredients;
2. Squamous cancer, small-cell lung cancer;
3. Symptomatic central nervous system (CNS) metastases
4. Hypertension and couldn't be controlled with medicine;
5. Coagulation disorders;
6. Clinical significant bleeding in 3 months prior dosing;
7. Had surgery in four weeks prior dosing;
8. Disease that affect drug absorption, such as inability to swallow, chronic diarrhea and intestinal obstruction;
9. Abdominal fistula, gastrointestinal perforation or intraperitoneal abscess in 6 months prior dosing;
10. Urine protein ≥++, and urine protein ≥1.0g in 24 hours;
11. Active infection and need antimicrobial treatments;
12. History of psychiatric substance abuse;
13. Take any clinical trial drugs within four weeks prior dosing;
14. Take any drugs that have effect on gastric acid and metabolic enzyme CYP 3A and CYP2D6;
15. Combined with other viral infections (anti-HCV, anti-HIV positive, HBsAg positive) or combined with syphilis infection;
16. Addicted to alcohol and tobacco;
17. Take grapefruit or grapefruit product, drinks containing caffeine, xanthine and alcohol in 48 hours prior dosing;
18. The investigator believes that the subjects are not eligible to participate in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2020-05-26 (Actual); Primary Completion 2021-02 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Cmax | 0-24 hours
  Maximum Observed Plasma Concentration for apatinib
AUC0-τ | 0-24 hours
  Area Under the Concentration-time Curve From Zero (Pre-dose) to 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-Sen Univercity Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Ma Y, Chen Q, Zhang Y, Xue J, Liu Q, Zhao Y, Yang Y, Huang Y, Fang W, Hou Z, Li S, Wang J, Zhang L, Zhao H. Pharmacokinetics, safety, tolerability, and feasibility of apatinib in combination with gefitinib in stage IIIB-IV EGFR-mutated non-squamous NSCLC: a drug-drug interaction study. Cancer Chemother Pharmacol. 2023 Nov;92(5):411-418. doi: 10.1007/s00280-023-04563-2. Epub 2023 Jul 31. PMID 37518060